CLINICAL TRIAL: NCT00417417
Title: Effects of Interleukin-1 Inhibition on C-Reactive Protein Levels, Endothelial Progenitor Cell Mobilization and Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Rilonacept to Improve Artery Function in Patients With Atherosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Richard Cannon, senior investigator, NHLBI Division of Inrtramural Research, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070055; 07-H-0055 (Other: NIH Clinical Center protocol 07-H-0055)
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Inflammation; Endothelial Dysfunction
Keywords: Endothelium; Inflammation; Nitric Oxide; Rilonacept; Cytokines; Coronary Artery Disease; CAD; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Inflammation | interventions — rilonacept; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rilonacept (Experimental): Rilonacept 320 mg subcutaneous at each treatment visit
  Interventions: Drug: Rilonacept
- Placebo (Sham Comparator): Normal saline subcutaneously at each treatment visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilonacept — Lyophilized rilonacept will be supplied by Regeneron Pharmaceuticals at 160 mg/vial and reconstituted with 2.3 mL of sterile water for injection by the Clinical Center Pharmacy Intravenous Admixture Unit. The formulation contains 80 mg/mL rilonacept, histidine, citrate, PEG 3350, polysorbate 20, glycine, arginine, and sucrose (pH 6.5). Matching placebo in the identical formulation will also be supplied, and also reconstituted with 2.3 mL of sterile water for injection. Each administration of study drug will consist of two syringes containing 2.0 mL in each syringe (320 mg total drug).
  Other Names: Arcalyst (brand name)
  Arms: Rilonacept
Drug: Placebo — Normal saline subcutaneously at each treatment visit.
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
This study will determine whether an experimental drug called Rilonacept can improve artery function in patients with atherosclerosis, a disease in which fatty deposits in arteries cause the vessels to stiffen, impeding blood flow. Atherosclerosis is believed to be caused in part by inflammation. Rilonacept blocks production of a protein called CRP, which, in high levels in the blood is associated with increased inflammation. Patients with coronary artery disease who have elevated blood levels of CRP are at increased risk of heart attack, heart failure and sudden death compared with people who have lower levels of the protein.

Patients 18 years of age and older with atherosclerotic coronary artery disease with a CRP level between 2 and 10 mg/L may be eligible for this study.

Patients are randomly assigned to receive four doses of either Rilonacept or placebo, given at 2-week intervals as injections under the skin. In addition to treatment, patients undergo the following procedures during eight visits to the NIH Clinical Center:

* Visit 1 (screening visit): Medical history, measurement of vital signs (temperature, blood pressure, heart rate and breathing rate), electrocardiogram (EKG) and blood tests.
* Visit 2: Blood tests, chest X-ray, treadmill exercise testing, tuberculin skin test, brachial artery flow-mediated dilation. Brachial artery flow-mediated dilation is used to measure how well the brachial artery (artery inside the elbow) dilates. An ultrasound device placed just above the elbow measures the size of the brachial artery and the flow of blood through it before and after a pressure cuff is inflated around the forearm.
* Visit 3: Injection of study drug.
* Visits 4, 5, and 6: Review of any changes in health or medical treatment, measurement of vital signs, blood tests, EKG, injection of study drug.
* Visit 7: Review of any changes in health or medical treatment, measurement of vital signs, blood tests, EKG, treadmill exercise testing, brachial artery flow-mediated dilation.
* Visit 8: Review of any changes in health or medical treatment, measurement of vital signs, blood tests, EKG, treadmill exercise testing, brachial artery flow-mediated dilation.

DETAILED DESCRIPTION:
Rilonacept (Interleukin-1 Trap) has been developed as an antagonist of the cytokine IL-1 in the treatment of rheumatoid arthritis and other inflammatory diseases. IL-1 causes leukocyte accumulation by inducing adhesion receptors on vascular endothelium and stimulating chemokine production. It also stimulates the synthesis of other cytokines, including IL-6, which in turn stimulates synthesis of C-reactive protein (CRP) in the liver. Based on numerous clinical studies, CRP has emerged as a risk marker for the development and clinical expression of atherosclerotic cardiovascular disease, leading to published recommendations for measurement of CRP in screening population subsets for cardiovascular risk. Endothelial function, as evidenced by stimulated nitric oxide release, has also been recognized as a marker of cardiovascular disease risk. Thus, patients with coronary artery disease (CAD) or its risk factors have impaired nitric oxide release from the endothelium compared with healthy subjects. Recent studies have shown that CRP levels were significantly higher in CAD patients compared with healthy subjects, with an inverse correlation between forearm blood flow responses to acetylcholine as a measure of endothelial function and CRP. Endothelial progenitor cells (EPCs) are primitive bone marrow-derived cells that have a capacity to home to sites of vascular injury and differentiate into vascular cell types, and are reduced in number and differentiation capacity in CAD patients relative to healthy subjects. Studies suggest that CRP inhibits viability and endothelial differentiation capacity of EPCs and may account for reduced numbers of EPCs and endothelial dysfunction in CAD patients. The objective of the present study is to demonstrate the potential of an investigational biological agent, rilonacept, as adjunctive treatment for CAD by examining effects of this agent on CRP levels, endothelial progenitor cell mobilization and endothelial function in a randomized, double-blind, placebo-controlled phase I/II clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male and non-pregnant female subjects over 18 years of age
* Diagnosis of atherosclerotic CAD by coronary angiography
* High sensitivity C-reactive protein (hsCRP) between 2.0 and 10.0 g/L, inclusive with percent change in CRP from Visit 1 to Visit 2 of less than 50% to +100%.
* Taking a HMG-CoA reductase inhibitor -For men and women of childbearing potential, willingness to utilize adequate contraception
* Willing, at time of study enrollment, to return for all clinic visits specified in the protocol and complete all study-related procedures.

EXCLUSION CRITERIA:

* BMI (body mass index) greater than 49.9 kg/m2 at Screening Visit 1 -Vascular intervention within 60 days prior to Screening Visit 1.
* Infection, use of systemic antibiotics, or clinically significant trauma (including surgery) within 30 days prior to Screening Visit 1.
* History or evidence of acute coronary syndrome within 60 days prior to Screening Visit 1.
* Acute or chronic inflammatory condition other than atherosclerosis
* Recently diagnosed diabetes mellitus
* Clinical evidence of congestive heart failure NYHA Class III-IV
* History of hypersensitivity other than localized injection site reaction to any biologic agent.
* Use of a thiazolidinedione
* Use of immunosuppressive or immunomodulatory medication (use of an inhaled glucocorticoid is permitted).
* Prior use of an immunomodulatory biologic drug within the last 6 months except immunizations and biologics used as standard care in cardiac care settings.
* Received a live/live attenuated vaccine within 90 days prior to Screening Visit 1 or other immunization within 30 days prior to Screening Visit 1.
* Prior or planned organ transplant recipient.
* Severe respiratory disease
* A history of tuberculosis infection, history of a positive skin test for tuberculosis, or a chest radiograph at Screening Visit 1 consistent with prior tuberculosis infection
* Positive result (5 mm or more in duration at 48 to 72 hours post-placement) of the PPD 5 TU placed at Screening Visit 2
* History or presence of malignancy (except for successfully treated basal cell carcinoma of the skin or in situ carcinoma of the cervix) within the past 5 years.
* HIV positive.
* Hepatitis B surface antigen or Hepatitis C antibody positive
* ALT, AST or alkaline phosphatase greater than twice the upper limit of the normal range, serum creatinine or total bilirubin greater than 1.5 times the upper limit of normal at Screening Visit 1.
* Hemoglobin less than 11.0 gm/dL, white blood cell (WBC) count less than 3,000/mm3, neutrophil count less than 2000/mm3 or platelet count less than 100,000/mm3 at Screening Visit 1.
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days prior to Screening Visit 1.
* History of substance abuse
* Elective surgery or vascular intervention planned to occur during the study.
* Any medical condition which would interfere with participation in the study, interfere with interpretation of study outcome measures, or place the subject at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard O Cannon, MD, Principal Investigator — NHLBI, NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dinarello CA. Biologic basis for interleukin-1 in disease. Blood. 1996 Mar 15;87(6):2095-147. PMID 8630372
- [Background] Colotta F, Re F, Muzio M, Bertini R, Polentarutti N, Sironi M, Giri JG, Dower SK, Sims JE, Mantovani A. Interleukin-1 type II receptor: a decoy target for IL-1 that is regulated by IL-4. Science. 1993 Jul 23;261(5120):472-5. doi: 10.1126/science.8332913.
- [Background] Dinarello CA. Interleukin 1 and interleukin 18 as mediators of inflammation and the aging process. Am J Clin Nutr. 2006 Feb;83(2):447S-455S. doi: 10.1093/ajcn/83.2.447S. PMID 16470011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with coronary artery disease were recruited from the Clinical Center outpatient clinic, and began in January, 2007.
Groups:
- Rilonacept: rilonacept 320 mg injected every 2 weeks x4 administrations.
- Placebo: placebo injected every two weeks x 4 administrations
Period: Overall Study
Arm/Group | Rilonacept | Placebo
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: placebo injected every two weeks for two months
- Total: Total of all reporting groups
Arm/Group | Rilonacept | Placebo | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (11) | 71 (10) | 69 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10
C-reactive protein [Mean (Standard Deviation); unit: mg/L] | 3.6 (1.8) | 3.9 (1.1) | 3.8 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: C-Reactive Protein (CRP)
Description: C-reactive protein levels in subjects randomized to rilonacept versus placebo injections.
Time Frame: 2 wks following last drug administration
Population: per protocol
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Rilonacept: rilonacept 320 mg x 4 administrations over 8 weeks.
- Placebo: Placebo x 4 injections over 8 weeks
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 4 | 6
mg/L | 3.7 (3.6) | 4.6 (2.7)

2. Other Pre Specified Outcome: Brachial Artery Flow-mediated Dilation
Description: Brachial artery flow-mediated dilation in respone to 5 minutes of forearm ischemia
Time Frame: Two weeks following final administration of drug
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Rilonacept: Rilonacept 320 mg subcutaneously x4 over 8 weeks
- Placebo: Placebo subcutaneous injection x 4 over 8 weeks
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 4 | 6
percent change | 6.3 (4.8) | 6.5 (3.6)

ADVERSE EVENTS:
Time Frame: Two years.
Description: 81 year-old man experienced viral upper respiratory infection following the second injection of the study drug. Because of rapid resolution of symptoms, he continued to receive the final two study injections, without incident. This adverse event was reported to the DSMB, the IRB, the FDA and Regeneron on April 16, 2007.
Arm/Group | Rilonacept | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rilonacept (N=4) | Placebo (N=6)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 81 year-old man who experienced viral upper respiratory infection following the second injection of placebo. Because of rapid resolution of symptoms, he continued to receive the final two study injections, without incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No